CLINICAL TRIAL: NCT03269487
Title: PERFECTED WP2: Implementing the Optimisation of Hospital Care Delivery to Older Adults by NHS Staff Via Action Research
Brief Title: PERFECTED WP2: Implementing Optimised Hospital Care
Acronym: PERFECTED
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: v1 01.04.2015
Record Dates: First submitted 2017-08-01; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2015-05

CONDITIONS: Implementation of Enhanced Recovery Pathway

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthcare professionals in partner sites: NHS employee or student nurse involved in the delivery of care to patients on partner wards in which the PERFECTED ERP is being implemented.

SUMMARY:
This study is part of the 5-year long (2013-18) PERFECTED (Peri-operative Enhanced Recovery hip-fracture Care of paTiEnts with Dementia) National Institute for Health Research (NIHR) funded research programme.

PERFECTED's aim is to develop and pilot an evidence-based intervention to improve the hospital care of patients living with dementia who have fractured their hip. This protocol relates to Work Package 2 (WP2) of PERFECTED only.

By working collaboratively with local clinicians and stakeholders, an action research (plan-do-study-act) approach will be used to generate knowledge to understand how to best implement the intervention (PERFECTED Enhanced Recovery Pathway), which was developed from learning and research undertaken as part of Work Package 1. During the current study the PERFECTED Enhanced Recovery Pathway (ERP) will be used to optimise care on three ortho-geriatric wards for 12 months. These wards are located in Norfolk, Nottinghamshire and Yorkshire. The sole participants are NHS personnel delivering care on selected wards.

Data collection activities (observations, in-field interviews, documentary analysis and quantitative data generated from the PERFECTED ERP implementation checklist) will determine the staff training and cultural changes required to implement and maximise adherence to the PERFECTED ERP. Simultaneously, enabling the identification and exploration of areas of optimised, satisfactory and sub-optimal care. By working in partnership within and across the partner wards, action plans to address sub-optimal care will be generated, implemented and reviewed. Findings will inform the best ways to optimise care via the implementation of the PERFECTED ERP. Knowledge generated during this study will be used to develop an ERP and staff training manual. This will aid implementation of the intervention arm of a latter Cluster Randomised Control Trial (Work Package 3), ensuring the PERFECTED ERP can be utilised in the real world.

As part of PERFECTED's commitment to Public Patient Involvement (PPI), lay researchers will be trained to assist with qualitative research activities.

ELIGIBILITY:
Inclusion Criteria:

* NHS employee or student nurse
* Involved in the delivery of care to patients on partner wards in which the PERFECTED ERP is being implemented

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sole participant group for this study are NHS employees involved in care delivery on partner hospital wards.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
PERFECT-ER | 12 months
  Improvement toolkit